CLINICAL TRIAL: NCT05946824
Title: Daily-Adaptive Stereotactic Body Radiation Therapy for Biochemically Recurrent, Radiologic Apparent Prostate Cancer After Radical Prostatectomy
Brief Title: This Study is Evaluating a New Radiation Treatment Technique for Patients Who Have Had Prostate Cancer, Undergone Surgery for Cancer, and Then Have Evidence That Their Prostate Cancer Has Returned.
Acronym: DASBRT-RPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Michael Cummings, Michael Andrew Cummings, M.D., Assistant Professor of Radiation Oncology, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URGUP22037
Record Dates: First submitted 2023-06-06; First posted 2023-07-14 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Prostate Cancer After Surgery
Keywords: Stereotactic body radiation therapy; daily-adaptive radiation therapy; prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This will be a two cohort Phase II single center, prospective trial, with a safety lead-in component. The cohorts will be defined by location of recurrence - either prostate bed alone, or a pelvic node with or without a prostate bed recurrence. This design will allow an initial toxicity assessment phase of a novel radiation treatment schema that is based on other literature, but with limited evidence. There is no plan to escalate the dose. Pending assessment of the safety lead in, complete enrollment will be permitted. Each cohort will be analyzed separated for the safety lead in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1 - Prostate bed only recurrence (Experimental): Patients with confirmed radiologic recurrence of their prostate cancer in the defined region of the previous prostate surgery - commonly referred to as the prostate surgical bed.
  Interventions: Radiation: Daily-adaptive Stereotactic Body Radiation Therapy
- 2- Pelvic nodal with or without a prostate bed recurrence (Experimental): Patients who have a radiologic recurrence of prostate cancer in the pelvic node region
  Interventions: Radiation: Daily-adaptive Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Daily-adaptive Stereotactic Body Radiation Therapy — Daily-adaptive radiation therapy to two dose levels - one to the area of radiologic recurrent nodal disease, and a lower, prophylactic dose to the standard post-prostatectomy and larger pelvic node fields
  Arms: 1 - Prostate bed only recurrence
Radiation: Daily-adaptive Stereotactic Body Radiation Therapy — Daily-adaptive radiation therapy to two areas - a high dose to the area of radiologic recurrence, and a lower, prophylactic dose to the standard post-prostatectomy fields
  Arms: 2- Pelvic nodal with or without a prostate bed recurrence

SUMMARY:
There is significant, proven use of radiation for recurrent prostate cancer after surgical resection. This treatment typically is delivered over seven and a half weeks of daily treatments, presenting a burden to patients and the health care system. Stereotactic body radiation (SBRT) is a radiation technique in which large doses are delivered over a short period of time. To date there is extremely limited evidence in SBRT for recurrent prostate cancer after surgery, with a significantly growing body of evidence for primary SBRT treatment of prostate cancer in men who opt for non-surgical upfront treatment. Additionally, advances in imaging have allowed better detection of the site of recurrence, and novel artificial intelligence aided daily-adaptive radiation therapy have allowed more precise delivery of radiation doses. This study seeks to evaluate the role of Daily-Adaptive with AI-assisted SBRT in the post operative setting utilizing Ethos Plan Adaptive technology in attempt to maintain control and minimize side effects.

DETAILED DESCRIPTION:
This will be a two cohort Phase II single center, prospective trial, with a safety lead-in component. This design will allow an initial toxicity assessment phase of a novel radiation treatment schema that is based on other literature, but with limited evidence. There is no plan to escalate the dose. Pending assessment of the safety lead in, complete enrollment will be permitted. Each cohort will be analyzed separated for the safety lead in. There will be 7 patients in the safety lead in cohorts. The stopping point will be an incidence of 2 cases of CTCAE v5.0 Grade 3+ acute toxicity attributed to therapy within gastrointestinal or urinary domains. This generally entails symptoms significant enough to require a procedure or limit basic levels of daily activity (bathing, cooking). Actue toxicity of a comparable magnitude has been reported in the 1-5% rate in a recent meta-analysis of contemporary trials which utilized standard of care radiation. Thus two cases would represent an unacceptable increased toxicity level, and a cohort size of 7 is approximate the commonly accepted size in Phase I escalation studies to evaluate dose limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate with previous surgical resection
* Radiologically detected prostate bed OR regional nodal recurrence defined as iliac, obturator, perirectal or pre-sacral node generally encompassing below the aortic bifurcation
* Prostate bed recurrence as occurring within the region of the prostate or RTOG consensus definition of the surgical field
* At least two serum detectable PSA levels defined as >0.02 ng/dl at least 30 days apart.

Exclusion Criteria:

* Metastatic disease
* Prior radiation therapy to the pelvis region
* Inflammatory bowel disease
* Hospitalization for a gastrointestinal diagnosis in the preceeding 3 months
* Hospitalization for a urinary tract issue / diagnosis in the preceeding 3 months
* PSA >10 ng/dl at study entry,

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must have prostate cancer to be eligible
Enrollment: 80 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2028-11-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | 1-2 years
  The Primary objective of the safety lead in component is to report acute, attributable genitourinary and gastrointestinal toxicity as scored by CTCAE v5.0.
The primary objective of the full enrollment Phase II component is to report biochemical recurrence free survival (bPFS). | 5 years
  We will utilize a globally standard definition of bPFS which was defined in the RADICALS(6) international trial as follows: freedom from PSA of 0·4 ng/mL or greater following postoperative radiotherapy, or PSA of more than 2·0 ng/mL at any time following therapy, clinical progression, or initiation of non-protocol hormone therapy, or death from any cause.

SECONDARY OUTCOMES:
Long term side effects | 5 years
  Late patient toxicity as defined by EPIC-IPSS prostate QoL forms
Distant metastasis free survival | 5 years
  Development of metastatic prostate cancer to other parts of the body
Need for long term anti-testosterone therapy | 5 years
  Time to initiation of non-protocol hormonal therapy, if needed

OTHER OUTCOMES:
Planning parameters and techniques | 5 years
  Identification of novel artificial-intelligence aided planning techniques, algorithms, and utilization as uncovered during the course of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmot Cancer Institute - Dept of Radiation Oncology, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided